CLINICAL TRIAL: NCT01412229
Title: A Phase II Study of Carboplatin, Nab-paclitaxel and Cetuximab for Induction Chemotherapy for Locally Advanced Squamous Cell Carcinoma of the Head and Neck
Brief Title: Induction Chemotherapy for Locally Advanced Squamous Cell Carcinoma of the Head and Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC1103
Record Dates: First submitted 2011-08-05; First posted 2011-08-09 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-09

CONDITIONS: Head and Neck Cancer
Keywords: Head and neck cancer; Phase II; Locally advanced; Squamous Cell; Carboplatin; Nab-paclitaxel; Abraxane; Cetuximab; Induction; Chemotherapy
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Cetuximab; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): * nab-paclitaxel 100mg/m2
  * Carboplatin area under curve (AUC)2 (IV)
  * Cetuximab 400mg/m2 week 1 then 250mg/m2 for six weeks
  Interventions: Drug: Cetuximab; Drug: Nab-paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Cetuximab — Weekly cetuximab given intravenously for 6 weeks during induction chemotherapy and continue during the 2-3 week break prior to definitive chemoradiotherapy.
  Other Names: Erbitux
Drug: Nab-paclitaxel — Weekly nab-paclitaxel given intravenously following cetuximab infusion for 6 weeks.
  Other Names: Abraxane
Drug: Carboplatin — Weekly carboplatin given intravenously following nab-paclitaxel infusion for 6 weeks.
  Other Names: Paraplatin

SUMMARY:
This is a non-randomized, open-label phase II trial of 40 patients with poor prognosis head and neck cancer, defined as surgically unresectable and/or ≥N2b disease and judged appropriate for non-surgical definitive therapy.

DETAILED DESCRIPTION:
This is a non-randomized, open-label phase II trial of 40 patients with poor prognosis head and neck cancer, defined as surgically unresectable and/or ≥N2b disease and judged appropriate for non-surgical definitive therapy. Patients must have Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 with good organ function and will be treated with six weekly cycles of carboplatin, nab-paclitaxel and cetuximab prior to scheduled concomitant chemoradiation. The study is designed to evaluate whether this induction regimen can result in an improved response rate (complete response (CR) + partial response (PR)) with less toxicity than the current standard induction docetaxel, cisplatin and 5-fluorouracil (TPF) regimen.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed SCCHN or poorly differentiated or undifferentiated cancer of the head and neck.
* Measurable disease.
* All primary sites are eligible excluding nasopharyngeal.
* Surgically unresectable and/or N2b or greater nodal disease; Note: surgical unresectability will be defined as the combination of the treating surgeon's judgment of unresectability plus one of the following objective criteria:

  * Encasement of tumor or nodes to the carotid artery or ¾ encasement of the carotid artery.
  * Involvement of prevertebral musculature
  * Invasion of the bone of the skull base
  * Need for glossectomy or extensive glossal resection where functional outcome is considered unacceptable to surgeon or patient
  * Involvement of the cervical spine
  * Severe, unacceptable functional deficit that would result from any proposed definitive surgical resection.
* ECOG performance status 0-1
* Prior therapy:

  * Chemotherapy: No prior chemotherapy for the treatment of SCCHN.
  * Platinum chemotherapy: No previous history of carboplatin or cisplatin therapy.
  * Nab-paclitaxel: No previous treatment with nab-paclitaxel or another taxane.
  * Cetuximab: No previous treatment with cetuximab Or another epidermal growth factor receptor (EGFR) inhibitor.
  * Radiation therapy: No prior radiation to the head and neck region.
* Age > or = 18 years. Men and women are eligible for participation.
* Must have acceptable organ and marrow function as defined below. Laboratory tests should be completed within 14 days prior to registration:

  * Absolute Neutrophil Count (ANC) > or = 1,500/mm3
  * Platelets > or = 100,000/mm3
  * Hemoglobin (Hgb) > 9g/dL
  * Total bilirubin < or = 1.5mg/dL
  * Albumin > 2.5 g/dL
  * Aspartate aminotransferase (AST)/Alanine Aminotransferase (ALT) < or = 2.5 times institutional upper limit of normal, alkaline phosphatase < 2.5 x upper limit of normal, glomerular filtration rate (GFR) > 30 mL/min (by standard Cockcroft and Gault formula or measured via 24 hour urine collection)
* No pre-existing neuropathy greater than grade I
* Women of childbearing potential must have a negative serum or urine pregnancy test performed within 7 days prior to day 1 of study treatment.
* Women of childbearing potential and men must agree to use adequate contraception prior to study entry, for the duration of study participation and for three months after completing treatment. Adequate contraception is defined as any medically recommended method (or combination of methods) as per standard of care.
* Patients must have the ability to understand and the willingness to sign a written informed consent document.
* Patients must have a negative result for preformed immunoglobulin E (IgE) antibodies to galactose-alpha-1,3,-galactose.

Exclusion Criteria:

* Prior treatment with any of the study medications.
* Prior radiation to any of the field required to treat the tumor.
* Any metastatic disease.
* The patient may have had a prior malignancy but must be disease-free for three years prior to study entry. A history of superficial non-melanoma skin cancer or in situ carcinoma of the cervix less than three years will be allowed.
* Pregnant or lactating female
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring IV antibiotics, or psychiatric illness/social situations that would limit compliance with study requirements. Cardiac disease such as symptomatic congestive heart failure, unstable angina pectoris, or myocardial infarction will result in exclusion only if active within the past six months. Cardiac dysrhythmia will only result in exclusion if active and symptomatic (for example, rate-controlled atrial fibrillation will not result in exclusion).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-02; Primary Completion 2015-06-20 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jared Weiss, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (3):
- United States (3):
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Vanderbilt University, Nashville, Tennessee
  - University of Washington, Seattle, Washington

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Homepage — http://unclineberger.org
- See also: National Cancer Institute Homepage — http://www.cancer.gov

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 10/12/2011 through 4/24/2015.
Pre-assignment Details: Sixty-seven subjects were consented to this trial. Of these, 29 were not eligible. 38 subjects were treated.
Groups:
- Treatment: * nab-paclitaxel 100mg/m2
  * Carboplatin Area under the Curve (AUC2) (IV)
  * Cetuximab 400mg/m2 week 1 then 250mg/m2 for six weeks
  Cetuximab: Weekly cetuximab given intravenously for 6 weeks during induction chemotherapy and continue during the 2-3 week break prior to definitive chemoradiotherapy.
  Nab-paclitaxel: Weekly nab-paclitaxel given intravenously following cetuximab infusion for 6 weeks.
  Carboplatin: Weekly carboplatin given intravenously following nab-paclitaxel infusion for 6 weeks.
Period: Overall Study
Arm/Group | Treatment
Started | 39
Completed | 38
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- Treatment: * nab-paclitaxel 100mg/m2
  * Carboplatin AUC2 (IV)
  * Cetuximab 400mg/m2 week 1 then 250mg/m2 for six weeks
  Cetuximab: Weekly cetuximab given intravenously for 6 weeks during induction chemotherapy and continue during the 2-3 week break prior to definitive chemoradiotherapy.
  Nab-paclitaxel: Weekly nab-paclitaxel given intravenously following cetuximab infusion for 6 weeks.
  Carboplatin: Weekly carboplatin given intravenously following nab-paclitaxel infusion for 6 weeks.
Arm/Group | Treatment
Number analyzed (Participants) | 39
Age, Continuous [Median (Full Range); unit: years] | 62 [46 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 32
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response Rate Following Induction Chemotherapy
Description: Evaluation of target lesions via imaging with CT or MRI scans at 2-3 weeks post induction chemotherapy. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions.
Time Frame: 9 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 39
Participants
  CR | 10
  PR | 20
  SD | 9

2. Secondary Outcome: Rate of Complete Response Following Induction Chemotherapy
Description: Report the rate of complete responses, defined as disappearance of all target lesions, following induction chemotherapy. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions.
Time Frame: Baseline evaluation to 3 weeks after induction chemotherapy
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 39
Participants | 10

3. Secondary Outcome: Progression Free Survival
Description: Rate of Progression Free Survival (Time to death or progression defined by imaging of target lesions via CT or MRI scan post induction chemotherapy and chemoradiotherapy every 3 months for one year)
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 39
percentage of participants | 81 [64 to 90]

4. Secondary Outcome: Objective Response Rate (CR+PR)
Description: Objective Response Rate as defined by RECIST 1.1 after induction chemotherapy followed by definitive chemoradiation. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Objective Response (OR) = CR + PR.
Time Frame: 20 weeks
Population: Patients who completed treatment
Measure: Count of Participants; unit: Participants
Groups:
- Treatment: * nab-paclitaxel 100mg/m2
  * Carboplatin area under curve (AUC)2 (IV)
  * Cetuximab 400mg/m2 week 1 then 250mg/m2 for six weeks
  Cetuximab: Weekly cetuximab given intravenously for 6 weeks during induction chemotherapy and continue during the 2-3 week break prior to definitive chemoradiotherapy.
  Nab-paclitaxel: Weekly nab-paclitaxel given intravenously following cetuximab infusion for 6 weeks.
  Carboplatin: Weekly carboplatin given intravenously following nab-paclitaxel infusion for 6 weeks.
Arm/Group | Treatment
Number analyzed (Participants) | 38
Participants | 30

5. Secondary Outcome: Complete Response Rate (CR)
Description: Complete Response Rate as defined by RECIST 1.1 after induction chemotherapy followed by definitive chemoradiation
Time Frame: 20 weeks
Population: Patients who completed treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 38
Participants | 10

6. Secondary Outcome: Overall Survival
Description: Rate of Overall Survival
Time Frame: 1 year
Population: Patients who completed treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 38
Participants | 34

7. Secondary Outcome: Number of Participants With at Least One Grade 3-4 Toxicity
Description: Toxicity will be assessed according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.
Time Frame: 9 Weeks
Population: Patients who received treatment on study
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 38
Participants | 17

8. Secondary Outcome: Number of Participants With at Least One Grade 3-4 Toxicity, Listed by Event
Description: as for outcome 7
Time Frame: 24 Weeks
Population: Patients who received study treatment
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 38
participants
  rash | 11
  decreased neutrophil count | 4
  decreased white blood cells | 2
  fatigue | 1
  palmar-plantar erythrodysesthesia syndrome | 1
  febrile neutropenia | 1
  hypocalcemia | 1
  hypokalemia | 1
  anaphylaxis to C225 | 0

9. Secondary Outcome: Patient-reported Quality of Life Scores
Description: Functional Assessment of Cancer Therapy - Head & Neck (FACT-HN) is the FACT-G and a 12 item head and neck cancer specific subscale completed at screening (Screening), 3 weeks post induction chemotherapy (Treatment Break), 7 weeks post concomitant chemoradiotherapy (7 weeks Off Treatment), one year post off-treatment (1 year Off Treatment). The FACT-G is a 27 item measure of general QOL assessing function in 4 domains: physical well-being (PWB), social-family well-being (SFWB), emotional well-being (EWB) and functional well-being (FWB). Items are rated by patients on a Likert scale from 0 to 4 (resulting in potential total scores between 0 and 156). Higher scores represent better QOL.
Time Frame: screening until one year after treatment
Population: All patients on treatment who returned completed questionnaires at each time point
Measure: Median (Full Range); unit: FACT-HN score
Arm/Group | Treatment
Number analyzed (Participants) | 36
FACT-HN score
  Pre-Treatment | 105.67 [43.33 to 142.00]
  Treatment Break: number analyzed (Participants) | 25
  Treatment Break | 117.00 [49.20 to 142.00]
  7 weeks Off Treatment: number analyzed (Participants) | 29
  7 weeks Off Treatment | 94.00 [58.00 to 132.00]
  1 year Off Treatment: number analyzed (Participants) | 22
  1 year Off Treatment | 116.00 [53.80 to 146.00]

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 13/39
Other Adverse Events (participants affected / at risk) | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=39)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Gallbladder obstruction (Hepatobiliary disorders) | 1 (1)
Gallbladder pain (Hepatobiliary disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) — increased secretions in oropharynx
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 (1) — biliary drain
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) — Pneumonia
Mucositis oral (Gastrointestinal disorders) | 2 (3)
Neutrophil count decreased (Investigations) | 2 (2)
Oral pain (Gastrointestinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Tracheal obstruction (Injury, poisoning and procedural complications) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=39)
Alanine Aminotransferase Increased (Investigations) | 10
Alkaline Phosphatase Increased (Investigations) | 5
Alopecia (Skin and subcutaneous tissue disorders) | 7
Anemia (Blood and lymphatic system disorders) | 27
Anorexia (Metabolism and nutrition disorders) | 13
Anxiety (Psychiatric disorders) | 8
Aspartate Aminotransferase Increased (Investigations) | 5
Blood Bilirubin Increased (Investigations) | 4
Constipation (Gastrointestinal disorders) | 23
Creatinine Increased (Investigations) | 7
Dehydration (Metabolism and nutrition disorders) | 6
Depression (Psychiatric disorders) | 4
Dermatitis Radiation (Skin and subcutaneous tissue disorders) | 9
Diarrhea (Gastrointestinal disorders) | 12
Dry Mouth (Gastrointestinal disorders) | 7
Dysgeusia (Nervous system disorders) | 9
Dysphagia (Gastrointestinal disorders) | 9
Fatigue (General disorders) | 23
Gastrointestinal Disorders - Other, Specify (Gastrointestinal disorders) | 7 — odynophagia, polydipsia, hematemesis; tracheostomy displacement, peg tube displacement
General Disorders And Administration Site Conditions - Other, Specify (General disorders) | 5 — Temperature Dysregulation, Subtherapeutic dilantin level, Mouth/Throat pain, Increased oral secretions, pain to throat and oral cavity
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 7
Hypoalbuminemia (Metabolism and nutrition disorders) | 5
Hypocalcemia (Metabolism and nutrition disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 6
Hypomagnesemia (Metabolism and nutrition disorders) | 24
Hyponatremia (Metabolism and nutrition disorders) | 11
Insomnia (Psychiatric disorders) | 7
Lymphocyte Count Decreased (Investigations) | 8
Mucositis Oral (Gastrointestinal disorders) | 17
Nausea (Gastrointestinal disorders) | 22
Neutrophil Count Decreased (Investigations) | 25
Oral Pain (Gastrointestinal disorders) | 13
Pain (General disorders) | 14
Peripheral Sensory Neuropathy (Nervous system disorders) | 4
Platelet Count Decreased (Investigations) | 12
Rash Acneiform (Skin and subcutaneous tissue disorders) | 34
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 5
Skin And Subcutaneous Tissue Disorders - Other, Specify (Skin and subcutaneous tissue disorders) | 6 — Cellulitis at percutaneous endoscopic gastrostomy (PEG) site; fissures, excoriation at g tube site, Abdominal skin tear around CT tube, cuticle disorder
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 4
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9
Vomiting (Gastrointestinal disorders) | 14
Weight Loss (Investigations) | 6
White Blood Cell Decreased (Investigations) | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other